CLINICAL TRIAL: NCT04981964
Title: Effect of Forward Versus Backward Walking Training on Back Geometry and Mobility Function in Children With Cerebral Palsy: a Randomized Controlled Study
Brief Title: Altered Back Geometry and Mobility Function After Backward Walking Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Almaz Abdel-Aziem, Professor of Biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002802
Record Dates: First submitted 2021-06-25; First posted 2021-07-29 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy plus forward walking (Experimental): 25 minutes of the forward walking training program It is based on methods as described by Grecco et al. (2013) The children were instructed to walk at a comfortable, self-selected speed during the first and final five minutes of the session and encouraged to increase the speed during the other 15 minutes.
  Interventions: Procedure: Exercise training
- Conventional physical therapy plus backward walking (Experimental): 25minutes of the backward walking training It is based on methods as described by Davis (1992) Firstly, the subject is asked to take a step backwards within the parallel bar and can support him or herself with the unaffected hand as required. The therapist provides help to move the subject's leg in the correct pattern, preventing subject from moving the leg back in full extension, when the subject can move the leg back with the correct pattern, the therapist gradually reduces the amount of assistance. Secondly, as the movement components have been practiced and the subjects has taken over actively with only slight help, the therapist facilitates walking backward within the parallel bars. Thirdly, the subject walks backwards actively away from the parallel bars. Finally, the distance and speed of walking backwards is progressively increased.
  Interventions: Procedure: Exercise training

INTERVENTIONS:
Procedure: Exercise training — both groups received conventional physiotherapy training program, for one hour, three sessions per week, for three successive months, based on neurodevelopmental treatment, composed of approximation of the upper and lower limbs in a regular and rhythmic manner, facilitation of righting, equilibrium and protective reactions, training of postural stability and equal weight shift especially on the affected side, stretching, strengthening exercises for upper and lower limbs and back muscles

SUMMARY:
PURPOSE: To assess the effect of backward walking training on back geometry and mobility function in children with hemiparetic cerebral palsy through a comparative analysis with forward walking training.

BACKGROUND:

Spinal deformities are important orthopaedic problems among children with cerebral palsy. A detailed evaluation of all these areas when the child first arrives for treatment is essential. The majority of research in children with CP is focused on assessment and treatment of upper and lower extremities. In contrast, literature on trunk control in children with CP is scarce. Although proximal trunk control is a prerequisite for improving balance and weight symmetry, there is a lack of studies that reported the role of forward and backward walking training in treating the trunk for children with CP. Therefore, the purpose of this study will investigate the role of backward walking training in addition to conventional physiotherapy program on back geometry and mobility function in children with spastic hemiparetic cerebral palsy.

HYPOTHESES: The null hypothesis of this study could be stated as: There will be no statistically significant difference in back geometry and mobility function after adding backward walking training to conventional physical therapy program in spastic hemiparetic cerebral palsy children compared with forward walking training.

RESEARCH QUESTION: Do adding backward walking training to conventional physical therapy program improves back geometry and functional mobility in children with hemiparetic cerebral palsy?

DETAILED DESCRIPTION:
Introduction:

Cerebral palsy (CP) describes a group of permanent disorders of the development of movement and posture, causing activity limitation. It is the most common cause of physical disability during childhood that affects the child on several health dimensions including neuromuscular deficits, such as spasticity, muscle weakness, and decreased selective motor control, and secondary musculoskeletal problems such as bony malformations and contractures.

Trunk impairment is very common but an underscored feature of spastic CP that affects the upper and lower extremity motor functions as well. Impairments associated with the trunk seen in children with CP include but are not limited with decreased stability of the head and trunk, shoulder protraction, spinal curve deviations, and trunk muscle weakness. Inadequate control of trunk muscles leads to compensation of other muscles to maintain the upright posture. Inability of proximal stabilization and increased activation of extremity muscles during postural adjustments reduces their functionality during extremity movements.

Trunk control is the initial frame of reference for postural control; it involves stabilization through selective movements of the trunk. Although trunk control strategies vary depending on the task and the environment, all functional tasks require adequate trunk control. Without the trunk as a stable center, selective movements of the extremities and of the head are profoundly impaired. In children, trunk control ensures the acquisition of basic gross motor skills in order to develop the goal-directed activities that are essential for independent life at home and in the community.

Evaluation of the CP child's passive and active movement of the trunk is an essential part of the evaluation because mobility of the spine in all planes is necessary for correct alignment, smooth and asymmetric movements of the spine and for full range of motion of the extremities. The therapist must document any deviation from normal, note scoliosis, excessive kyphosis and lordosis and whether the curves are structural or functional.

The majority of research in children with CP is focused on assessment and treatment of upper and lower extremities. In contrast, literature on trunk control in children with CP is scarce. Although proximal trunk control is a prerequisite for improving balance and weight symmetry, there is a lack of studies that reported the role of forward and backward walking training in treating the trunk for children with CP.

Material and methods

Subjects:

A thirty-eight spastic hemiparetic cerebral palsied children of both sexes will participate in this study. The participants will be selected from the out-patient clinic of faculty of physical therapy, Cairo university. All participants will be selected according to the following inclusive criteria: Their age ranged from 5 to 7 years, with average height around one meter or more as it is the suitable height for Formetric measures (because the horizontal line which appears on the computer screen when the camera is ready for recording should be below the scapula to avoid the un-detection of the axillary points which will interfere with recording of the spinal image). They were able to stand alone independently and have the ability to walk both forward and backward over ground without an assistive device. They were able to understand and follow verbal command. They will be classified as I or II by gross motor function classification system (GMFCS). The degree of spasticity in the involved lower extremity according to Modified Ashworth Scale ranged between grades 1, 1+ and 2. Exclusion criteria for all participants will be neurological or orthopedic surgery in the last 12 months, uncontrolled seizure disorder, visual, auditory or perceptual problems and who had any experience of backward training before the trial. This study protocol was approved by the research ethical committee of the Faculty of Physical Therapy, Cairo University (P.T.REC/012/002802) and parents will sign a consent form authorizing the child's participation.

The participants will be randomly allocated into 2 groups (group A and B). The participants of group (A) will receive physical therapy program based on neurodevelopmental treatment (NDT) approach, in addition a specially designed forward walking training program. The participants of group (B) will receive the same physical therapy program, in addition a specially designed backward walking training program.

For evaluation:

The assessment will be conducted for each child of both groups individually before and after three successive months of treatment by the same examiner who will be blinded to treatment allocation. The outcome measures will be;

1. Formetric instrument system
2. Dynamic Gait Index (DGI)

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 5 to 7 years
* Average height around one meter or more as it is the suitable height for formetric measures
* They were able to stand alone independently and have the ability to walk both forward and backward over ground without an assistive device.
* They were able to understand and follow verbal command. They were classified as I or II by gross motor function classification system (GMFCS).
* The degree of spasticity in the involved lower extremity according to Modified Ashworth Scale ranged between grades 1, 1+ and 2.

Exclusion Criteria:

* Neurological or orthopedic surgery in the last 12 months, uncontrolled seizure disorder, visual, auditory or perceptual problems and who had any experience of backward training before the trial.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Trunk imbalance | Change from Baseline Trunk imbalance at 3 months
  It represented the lateral deviation of the vertebra prominence from the dimple midpoint. It is measured in millimeters.
Lateral deviation | Change from Baseline Lateral deviation at 3 months
  The root mean square (RMS) lateral deviation of the spinal midline from the line VP-DM. It is measured in millimeters
Pelvic tilt | Change from Baseline Pelvic tilt at 3 months
  The pelvic tilt refers to a height difference of the lumber dimples relative to a horizontal plane. It is measured in millimeters
Surface rotation | Change from Baseline Surface rotation at 3 months
  The root mean square (RMS) value of the surface rotation on the symmetry line (in degrees).
Pelvic torsion | Change from Baseline Pelvic torsion at 3 months
  It is the twisting of the pelvis about a transverse axis (in degrees).

SECONDARY OUTCOMES:
Mobility function | Change from Baseline dynamic gait index at 3 months
  The Dynamic Gait Index (DGI) will be used to measure mobility function and dynamic balance in walking and stair climbing. There are 8 items on the DGI and each item is scored on a 4-point scale [(3) Normal; (2) Mild impairment; (1) Moderate impairment; (0) Severe impairment] with a maximal score of 24. The 8 items include walking, walking with speed changes, walking with vertical and then horizontal head turns, walking with a quick pivot stop, walking over objects, walking around objects and walking up and down stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Abdel-aziem, Ph.D, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, None Selected, Egypt